CLINICAL TRIAL: NCT02831010
Title: A Multi-Center Cohort Study of Risk Factors and Outcomes of Encephalopathy of Prematurity in China
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: EKYYEOPMC
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Encephalopathy
Keywords: prematurity
MeSH Terms: conditions — Brain Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- encephalopathy of prematurity: infants with encephalopathy of prematurity showed on MRI at term-equivalent age
- no encephalopathy of prematurity: infants with no encephalopathy of prematurity showed on MRI at term-equivalent age

SUMMARY:
The purpose of this study is to explore the perinatal risk factors of encephalopathy of prematurity and the morbidity of the following neurodevelopmental impairments in preterm infants with gestational age <32 weeks in China.

DETAILED DESCRIPTION:
Recent years have witnessed an increase in survival of very or extremely low birth weight infants, with a corresponding increase of attention to encephalopathy of prematurity (EOP) and the following neurological disorders. Studies suggested that hypoxic-ischemic injury and perinatal infection might be the two main risk factors of EOP, including white matter injury, neuronal-axonal diseases and cerebellar hemorrhage, which have a strong impact on neurological outcomes. Sequelae like cerebral palsy or mental retardation become a burden to both the family and society. Therefore, the risk factors of brain injury become the critical issue of both Obstetrics and Neonatology. More importantly, little is known about the morbidity of neurodevelopmental impairment and its risk factors in China. Thus, the aim of our study is to explore the perinatal risk factors of encephalopathy of prematurity and the morbidity of the following neurodevelopmental impairments in preterm infants with gestational age <32 weeks in China.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with gestational age less than 32 weeks

Exclusion Criteria:

* major congenital malformations
* chromosomal disorders
* metabolic diseases

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonatal intensive-care units
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2014-04; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
developmental quotient (DQ) on the Gesell Developmental Schedules | 2 years
  Result of gross motor, fine motor, language and social test. DQ = Development Age / Chronological Age X 100

SECONDARY OUTCOMES:
brain injury showed on MRI | 36-40 weeks' postmenstrual age or before discharge
  signal abnormality in white matter, grey matter or cerebellum injury; periventricular leukomalacia; intracranial hemorrhage
morbidity of encephalopathy of prematurity | 36-40 weeks' postmenstrual age or before discharge
  white matter injury, grey matter injury, cerebellum injury on MRI
all cause mortality | 2 years
  Mortality that does not require judgments about the cause of death
neurodevelopment sequelae | 2 years
  including cerebral palsy, epilepsy, hearing loss, vision loss, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chen, PhD, MD, Study Director — Children's Hospital of Fudan University
Locations (14):
- China (14):
  - The First People's Hospital of Hefei, Hefei, Anhui
  - Xiamen Women's and Children's Health Centre, Xiamen, Fujian
  - People's Hospital of Zhangzhou, Zhangzhou, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhongshan Bo Ai Hospital, Zhongshan, Guangdong
  - Maternal and Child Health Hospital of Guiyang Province, Guiyang, Guizhou
  - Handan Central Hospital, Handan, Hebei
  - First Hospital of Jilin University, Changchun, Jilin
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Maternity and Children's Hospital, Xian, Shanxi
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Ningbo Women's and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volpe JJ. Encephalopathy of prematurity includes neuronal abnormalities. Pediatrics. 2005 Jul;116(1):221-5. doi: 10.1542/peds.2005-0191. No abstract available. PMID 15995055
- [Background] Groenendaal F, Termote JU, van der Heide-Jalving M, van Haastert IC, de Vries LS. Complications affecting preterm neonates from 1991 to 2006: what have we gained? Acta Paediatr. 2010 Mar;99(3):354-8. doi: 10.1111/j.1651-2227.2009.01648.x. Epub 2010 Jan 8. PMID 20064132
- [Background] Volpe JJ. Brain injury in premature infants: a complex amalgam of destructive and developmental disturbances. Lancet Neurol. 2009 Jan;8(1):110-24. doi: 10.1016/S1474-4422(08)70294-1. PMID 19081519
- [Background] Korzeniewski SJ, Romero R, Cortez J, Pappas A, Schwartz AG, Kim CJ, Kim JS, Kim YM, Yoon BH, Chaiworapongsa T, Hassan SS. A "multi-hit" model of neonatal white matter injury: cumulative contributions of chronic placental inflammation, acute fetal inflammation and postnatal inflammatory events. J Perinat Med. 2014 Nov;42(6):731-43. doi: 10.1515/jpm-2014-0250. PMID 25205706
- [Background] Sominsky L, Walker AK, Ong LK, Tynan RJ, Walker FR, Hodgson DM. Increased microglial activation in the rat brain following neonatal exposure to a bacterial mimetic. Behav Brain Res. 2012 Jan 1;226(1):351-6. doi: 10.1016/j.bbr.2011.08.038. Epub 2011 Sep 1. PMID 21907243
- [Background] Shatrov JG, Birch SCM, Lam LT, Quinlivan JA, McIntyre S, Mendz GL. Chorioamnionitis and cerebral palsy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):387-392. doi: 10.1097/AOG.0b013e3181e90046. PMID 20664400
- [Background] Howson CP, Kinney MV, McDougall L, Lawn JE; Born Too Soon Preterm Birth Action Group. Born too soon: preterm birth matters. Reprod Health. 2013;10 Suppl 1(Suppl 1):S1. doi: 10.1186/1742-4755-10-S1-S1. Epub 2013 Nov 15. PMID 24625113
- [Background] Hendson L, Russell L, Robertson CM, Liang Y, Chen Y, Abdalla A, Lacaze-Masmonteil T. Neonatal and neurodevelopmental outcomes of very low birth weight infants with histologic chorioamnionitis. J Pediatr. 2011 Mar;158(3):397-402. doi: 10.1016/j.jpeds.2010.09.010. Epub 2010 Oct 18. PMID 20961565
- [Background] Sato M, Nishimaki S, Yokota S, Seki K, Horiguchi H, An H, Ishida F, Fujita S, Ao K, Yatake H. Severity of chorioamnionitis and neonatal outcome. J Obstet Gynaecol Res. 2011 Oct;37(10):1313-9. doi: 10.1111/j.1447-0756.2010.01519.x. Epub 2011 May 3. PMID 21535310